CLINICAL TRIAL: NCT03709836
Title: Computed Tomography Angiography Prediction Score for Side Branch Occlusion in Coronary Bifurcation Intervention (CT-PRECISION)
Brief Title: Computed Tomography Angiography Prediction Score for Side Branch Occlusion
Acronym: CT-PRECISION
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: 2.43/III/16
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Coronary bifurcation lesion; Coronary angiography; Coronary computed tomography angiography; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lesions involving coronary bifurcations account for approximately 20% of all percutaneous coronary interventions (PCI). Revascularization within bifurcation sites remains technically challenging. While the most optimal interventional treatment strategy for bifurcation lesions is still debatable, side branch (SB) occlusion is one of the most serious procedural complications with prevalence rates over 7%.

Numerous mechanisms of the SB occlusion (e.g. plaque or carina shift, coronary artery dissection, thromboembolism, coronary artery spasm, etc) have been postulated. Regardless of the cause, loss of the SB is associated with increased risk of periprocedural mortality and myocardial infarction. Therefore, PCI involving coronary bifurcation mandates consideration of the risk of SB compromise. The CT-PRECISION (Computed Tomography angiography PREdiCtIon score for SIde branch Occlusion in coronary bifurcation interventioN) registry was designed to evaluate the application of coronary computed tomography angiography (coronary CTA) for the prediction of SB occlusion during percutaneous revascularization of bifurcation lesions. The main purpose of this single-center study is to develop a noninvasive CTA-based prediction tool to determine the procedural outcome of PCI in bifurcation lesions.

DETAILED DESCRIPTION:
Coronary CTA allows for precise and noninvasive evaluation of coronary bifurcation lesions. Pre-procedural planning for coronary revascularization using CTA provides detailed characterization of bifurcation anatomy and morphology including the spatial distribution of coronary plaque. To date there has been no compiled CTA-based prediction model for SB occlusion in coronary bifurcation intervention.

The CT-PRECISION registry is a retrospective observational cohort study of patients undergoing preprocedural coronary CTA before PCI involving coronary bifurcation lesions between January 2010 and July 2018. The study is designed to enroll 400 consecutive patients undergoing elective main vessel stenting with a provisional approach to the SB at a single high-volume PCI center.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for attempted PCI of a bifurcation lesion with a significant SB as part of their standard of care
* Initial stenting of the main branch with a provisional approach to the SB
* Performance of dual-source coronary CTA within 30 days before attempted PCI

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients undergoing preprocedural coronary CTA before attempted PCI involving coronary bifurcation with a significant SB. All consecutive patients meeting all inclusion criteria and no exclusion criteria will be included within the CT-PRECISION registry.
Sampling Method: Probability Sample
Enrollment: 363 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
SB occlusion | intraprocedural
  SB occlusion defined as a any decrease in Thrombolysis in Myocardial Infarction (TIMI) flow grade or the absence of flow in the SB after main vessel stenting

CONTACTS AND LOCATIONS:
Overall Officials: Adam D. Staruch, MD, Principal Investigator — Department of Interventional Cardiology, and Angiology, Institute of Cardiology, Warsaw, Poland; Maksymilian P. Opolski, MD, PhD, Study Chair — Department of Interventional Cardiology, and Angiology, Institute of Cardiology, Warsaw, Poland; Adam Witkowski, MD, PhD, Study Chair — Department of Interventional Cardiology, and Angiology, Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grodecki K, Cadet S, Staruch AD, Michalowska AM, Kepka C, Wolny R, Pregowski J, Kruk M, Debski M, Debski A, Michalowska I, Slomka PJ, Witkowski A, Dey D, Opolski MP. Noncalcified plaque burden quantified from coronary computed tomography angiography improves prediction of side branch occlusion after main vessel stenting in bifurcation lesions: results from the CT-PRECISION registry. Clin Res Cardiol. 2021 Jan;110(1):114-123. doi: 10.1007/s00392-020-01658-1. Epub 2020 May 8. PMID 32385529
- [Derived] Opolski MP, Grodecki K, Staruch AD, Michalowska AM, Kepka C, Wolny R, Knaapen P, Schumacher SP, Pregowski J, Kruk M, Debski M, Debski A, Michalowska I, Witkowski A. Accuracy of RESOLVE score derived from coronary computed tomography versus visual angiography to predict side branch occlusion in percutaneous bifurcation intervention. J Cardiovasc Comput Tomogr. 2020 May-Jun;14(3):258-265. doi: 10.1016/j.jcct.2019.11.007. Epub 2019 Nov 21. PMID 31806391